CLINICAL TRIAL: NCT01069835
Title: Epidemiological Study to Describe NSCLC Clinical Management Patterns in Central Eastern Europe and Russia. Lung-EPICLIN
Brief Title: Epidemiological Study to Describe Non Small Cell Lung Cancer (NSCLC) Clinical Management Patterns in Central Eastern Europe and Russia (Lung-EPICLIN)
Acronym: EPICLIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ORU-IRE-2009/1
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; EGFR mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin embedded tumour tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Non-small cell lung cancer patients

SUMMARY:
The overall aim of the study is:

To provide accurate and reliable information regarding NSCLC clinical management across Central Eastern European countries and Russia in order to detect unmet medical needs of this disease in terms of:

* Patient and hospital characteristics.
* Diagnostic and treatment approaches: initial and subsequent.
* Follow-up patterns in clinical management.
* Outcomes: symptoms, death, functionality, quality of life.
* Use of resources and burden on patients and health care systems. Addendum objective is to collect epidemiological data on EGFR mutation status (M+, M-) in the Russian population

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NSCLC diagnosis (e.g.bronchoscopic biopsy or FNAB), all stages, men and women, attending the responsible department of treating this type of patients for the first time between January 1st, 2010 and March 31st, 2010
* For Patient Reported Outcome (PRO) sub-sample: ability to read and write since they will be asked to participate in the PRO part of the study. Selection will not be based on the disease stage of each patient, in order to avoid a selection bias.
* Tumour tissue samples (in paraffin-embedded blocks) suitable for EGFR mutation testing available.

Exclusion Criteria:

* Mixed histology of small cell and non-small cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients from Oncological Dispensaries and Cancer Research Institutes
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To assess the differences in patient characteristics, disease stage (differentiating between non-advanced disease, locally advanced disease, metastatic disease), and in clinical management across Central Eastern European countries and Russia | 24 months

SECONDARY OUTCOMES:
To detect differences in clinical outcomes and related factors among countries | 24 months
To identify factors associated with clinical outcomes (patient, disease stage -see above- and clinical management related factors): predictive modelling for improved patient outcome | 24 months
To identify factors associated with the different levels of functional status and quality of life | 24 months
To compare the use of health care resources among countries | 24 months

CONTACTS AND LOCATIONS:
Locations (31):
- Russia (31):
  - Research Site, Barnaul, Altaiskiy Krai
  - Research Site, Birobidzhan, EAO
  - Research Site, Khabarovsk, Khabarovskiy Krai
  - Research Site, Khanty-Mansyisk, Khanty-Mansyiskyi AO
  - Research Site, Krasnodar, Krasnodarskiy Krai
  - Research Site, Vladivostok, Primorskiy Krai
  - Research Site, Kazan', Resp. of Tatarstan
  - Research Site, Yakutsk, Sakha
  - Research Site, Arkhangelsk
  - Research Site, Belgorod
  - Research Site, Blagoveshchensk
  - Research Site, Chita
  - Research Site, Engel's
  - Research Site, Irkutsk
  - Research Site, Kemerovo
  - Research Site, Khimki
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Oryol
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Tomsk
  - Research Site, Tula
  - Research Site, Volgograd
  - Research Site, Yuzno-Sakhalinsk
  - Research Site, Zhukovsky

REFERENCES:
- [Derived] Tjulandin S, Imyanitov E, Moiseyenko V, Ponomarenko D, Gurina L, Koroleva I, Karaseva V. Prospective cohort study of clinical characteristics and management patterns for patients with non-small-cell lung cancer in the Russian Federation: EPICLIN-Lung. Curr Med Res Opin. 2015 Jun;31(6):1117-27. doi: 10.1185/03007995.2015.1036015. Epub 2015 May 8. PMID 25867537
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1019&filename=CSR-NIS-ORU-IRE-2009-1.pdf
- See also: CSR-NIS-ORU-IRE-2009-1.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1019&filename=CSR-NIS-ORU-IRE-2009-1.pdf
- See also: NIS-ORU-IRE-20091EPICLIN-LUNG-FinalProtocol-CEERussia-08122009 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1019&filename=NIS-ORU-IRE-20091EPICLIN-LUNG-FinalProtocol-CEERussia-08122009.pdf